CLINICAL TRIAL: NCT06114342
Title: The Biological Specificity of Acupoints Between Major Depressive Disorder Patients and Healthy Controls: A Prospective, Assessor-blinded, Comparative Study
Brief Title: The Biological Specificity of Acupoints Between Major Depressive Disorder Patients and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Xiaomei Shao (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 2022ZX010-IP
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Acupoint; Biological specificity
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HC group: There were 50 healthy control participants in the HC group.
- MDD group: There were 84 MDD patients in the MDD group. 50 MDD subjects were enrolled at each acupoint for each test.

SUMMARY:
Evidence-based medicine suggests that acupuncture can improve major depressive disorder (MDD). However, the prevalent reliance on experiential acupoint selection lacks scientific underpinning. The investigators conducted a comparative study involving MDD patients and healthy subjects, employing modern techniques to discern biological specificity in MDD-related acupoints. Additionally, the investigators investigated potential correlations between acupoint biological specificity and MDD severity.

DETAILED DESCRIPTION:
A final total of 134 eligible subjects were included. Among them, 50 healthy subjects were assigned to the healthy control (HC) group and 84 MDD participants were assigned to the MDD group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the healthy control participants:

* provided a recent depression screening report, and be free of any cardiovascular, respiratory, digestive, urinary, hematological, endocrine, or neurological disease;
* 18 ≤ age ≤60 years, male or female;
* had clear consciousness and could communicate with others normally; - understand the full study protocol and have high adherence;
* signed the written informed consent.

Inclusion criteria for the MDD participants:

* consistent with the diagnosis of MDD in the International Classification of Diseases 10th Edition (ICD-10);
* 18 ≤ age ≤ 60, male or female;
* had clear consciousness and could communicate with others normally;
* understand the full study protocol and have high adherence;
* signed the written informed consent.

Exclusion Criteria:

* The exclusion criteria of the HC participants were as follows: (1) had serious primary diseases of cardiovascular diseases, liver diseases, kidney diseases, urinary diseases, and hematological diseases; (2) pregnant or lactating; (3) had scars, hyperpigmentation, red and swollen of the skin at the test site; (4) were participating in other trials; (5) had a mental illness, alcohol dependence, or a history of drug abuse. Exclusion criteria for the MDD participants: (1)-(4) same exclusion criteria as healthy subjects; (5) MDD caused by organic mental disorders, schizophrenia, bipolar disorder, psychoactive substances, and non-addictive substances; (6) had psychiatric disorders other than MDD; (7) with suicidal tendencies. In addition, IRT is not be performed on female subjects during their menstrual and ovulatory periods.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The diagnostic criteria of MDD were based on criteria proposed by the International Classification of Diseases 10th Edition (ICD-10). Healthy control participants were determined by a recent depression screening report for confirming their mental health conditions.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Temperature | Baseline
  Temperature of acupoints was measured by infrared thermography (IRT). IRT was not be performed on female subjects during their menstrual and ovulatory periods.
Pressure pain threshold | Baseline
  Pressure pain threshold was measured by pressure pain threshold gauge (PTG).

SECONDARY OUTCOMES:
The Hamilton Depression Scale-17 (HAMD-17) Scores | Baseline
  The HAMD scale is the most commonly used in the clinical assessment of depression, including 17 items. The higher the score, the more severe the depression. 0-6 means no depressive symptoms, 7-16 means mild depression, 17-24 was divided into moderate depression, and more than 25 was divided into severe depression.
The Patient Health Questionaire-9 Items (PHQ -9) | Baseline
  The PHQ-9 scale has a total of 9 questions, each with a score of 0-3 (none: 0; a few days: 1; more than half of the time: 2; almost every day: 3), with a total score of 0-27.
The Self-Rating Depression Scale (SDS) Scores | Baseline
  The standard score is the total of all scores multiplied by 1.25 to the nearest whole number on this scale, which has 20 questions. A standard score below 50 is normal; 53-62 is mild depression; 63-72 is moderate depression; 72 or more is severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No